CLINICAL TRIAL: NCT01534429
Title: Quantitative Sensory Testing and Neurophysiologic Analysis of Post-Herniorraphy Pain in Patients Undergoing Selective Neurectomy and Mesh Removal
Brief Title: Quantitative Sensory Testing and Analysis of Post Inguinal Hernia Surgery Pain
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 11-000180
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Hernia
Keywords: pain
MeSH Terms: conditions — Hernia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic post-herniorraphy pain: patients with severe chronic post-herniorraphy pain
  Interventions: Procedure: Quantitative Sensory Testing

INTERVENTIONS:
Procedure: Quantitative Sensory Testing — Quantitative Sensory Testing and Neurophysiologic Testing to be done Pre-operatively and at 3 and 6 months post-operatively.

SUMMARY:
Increasing experience has identified post-herniorraphy chronic pain as an under-recognized and important complication. Nerve entrapment and injury are recognized as causes of such pain. Operative treatment for selected patients with this condition includes surgical exploration of the affected groin, identification and removal of involved nerves, and removal of meshoma. This procedure has been highly effective in treatment of chronic pain. This study will attempt to subjectively and objectively evaluate the patient's chronic groin pain using quantitative sensory testing (QST) and validated pain scales and questionnaires. Quantitative sensory testing is a method used to assess damage to the small and large nerve fibers. It is used to diagnose and assess the severity of nerve damage, and can also help to determine if a neuropathy is responding to treatment. QST uses a computer testing system to measure how nerves react to vibration and changes in temperature. The procedure is non-invasive and the patient will feel minimal to no discomfort during testing. The hypothesis is that any decrease in subjective pain scores would be accompanied by improved QST results.

DETAILED DESCRIPTION:
Background: Chronic postherniorrhaphy inguinal pain is a complex, major health problem. In the absence of recurrence or meshoma, laparoscopic retroperitoneal triple neurectomy has emerged as an effective surgical treatment of postherniorrhaphy inguinal pain. Methods: This prospective pilot study evaluated the neurophysiological and clinical effects of laparoscopic retroperitoneal triple neurectomy. Ten consecutive adult with chronic postherniorrhaphy inguinal pain and unilateral predominantly neuropathic inguinodynia underwent three comprehensive quantitative sensory testing assessments (preoperative, immediate postoperative, and late postoperative). Pain severity, health-related function, and sleep quality were assessed over the course of a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* patient with chronic groin pain after inguinal hernia surgery and are candidates for triple neurectomy with mesh removal

Exclusion Criteria:

* non-English speaking patients
* significant psychiatric or medical disease
* bilateral groin pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain occuring after groin hernia repair who are surgical candidates for mesh removal and triple neurectomy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
changes in quantitative sensory testing and neurophysiologic testing pre-operatively, and at 3-month and 6-month intervals post-operatively | 6 months

SECONDARY OUTCOMES:
changes in Visual Nociceptive Pain Scores, McGill Pain Questionnaire, Activity Assessment Scale, and SF-36 scale pre-operatively and 3-month, 6-month, and 9-months post-operatively | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Nicol, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No